CLINICAL TRIAL: NCT06277427
Title: Refractory ANCA Associated Vasculitis and Lupus Nephritis Treated With BCMA-targeting CAR-T Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lingli Dong (Other)
Collaborators: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Lingli Dong, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]S208
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Lupus Nephritis; ANCA Associated Vasculitis
Keywords: CAR-T; Lupus nephritis; ANCA associated vasculitis; BCMA
MeSH Terms: conditions — Lupus Nephritis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment (Experimental): Lymphocyte clearance before PRG-1801 cells' infusion; Plan to design two dose levels (2.5x10^6 CAR-T/kg and 5.0x10^6 CAR-T/kg), with 3-6 AAV and LN subjects included in each dose group, totaling 12-24 subjects. Within each dose group, the next subject can be administered after the previous subject has completed at least 14 days of safety observation.
  Dose group 1: with a dosage of 2.5x10^6 (cells/kg) per dose Dose group 2: with a dosage of 5.0x10^6 (cells/kg) per dose
  Interventions: Drug: PRG-1801 （CAR-T against BCMA）

INTERVENTIONS:
Drug: PRG-1801 （CAR-T against BCMA） — Patients with refractory LN and ANCA-associated vasculitis will be treated with PRG-1801

SUMMARY:
Lupus nephritis (LN) and ANCA-associated vasculitis are severe autoimmune diseases, which may lead to the death of patients, particularly when they are refractory to the conventional therapeutic agents. Based on the current knowledge, the autoantibodies against self-antigens may exert important pathological roles in the pathogenesis of both LN and ANCA-associated vasculitis, of which the origins are primarily plasmablasts and plasma cells. BCMA is the molecule expressed on memory B cells, plasmablasts and plasma cells, and therefore is an ideal target for the elimination of potential pathogenic antibody secreting cells. Chimeric antigen receptor (CAR) T cells against BCMA may provide a novel therapeutic way for the refractory LN and ANCA-associated vasculitis patients to eliminate the pathogenic autoantibody-secreting cells. In this study, the safety and efficacy of a novel CAR-T cell therapy using PRG-1801 cells, are evaluated in patients with refractory LN and ANCA-associated vasculitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, not exceeding 70 years old (including 70 years old);
2. If the kidneys are involved, estimate the glomerular filtration rate (eGFR) to be ≥ 15 mL/minute/1.73 m2;
3. The following test values within 3 days before the collection of mononuclear cells meet the following standards:

   1. Absolute lymphocyte count: ≥ 0.5 × 10 ^ 9/L [The use of granulocyte colony-stimulating factor (G CSF) is allowed, but subjects are not allowed to receive this supportive treatment within 7 days before the screening period laboratory examination];
   2. Absolute neutrophil count: ≥ 1.0 × 10 ^ 9/L [The use of granulocyte colony-stimulating factor (G-CSF) is allowed, but subjects are not allowed to receive this supportive treatment within 7 days before the screening period laboratory examination];
   3. Platelets: Subject platelet count ≥ 50 × 10 ^ 9/L (subjects are not allowed to receive blood transfusion support within 7 days before the screening period laboratory examination);
   4. Hemoglobin: ≥ 8.0 g/dL (allowing the use of recombinant human erythropoietin) [subjects have not received red blood cell (RBC) infusion within 7 days prior to the screening period laboratory examination];
   5. Creatinine clearance rate: (CrCl) or glomerular filtration rate (GFR) (Cockcroft Gault formula) ≥ 30 mL/min;
   6. Total bilirubin (serum): Total bilirubin (serum) ≤ 1.5 × ULN; Blood bilirubin>1.5 × Gilbert subjects from ULN can be enrolled with the consent of the sponsor
   7. AST and ALT: ≤ 3.0 × ULN;
   8. Plasma prothrombin time (PT), international standardized ratio (INR), partial prothrombin time (APTT): PT ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN, INR ≤ 1.5 × ULN
4. Willing to sign an informed consent form.
5. - for refractory ANCA-associated vasculitis

   ①According to the 2022ACR/EULAR criteria, diagnosed with AAV (GPA or MPA subtype), who has not achieved remission (BVAS score of 0) for ≥ 3 months after receiving standardized treatment. Severe patients who have previously undergone standardized treatment to induce remission and are now relapsing after maintenance therapy; ②The patient is currently or has a positive ANCA during the course of the disease; ③Severe illness (severe organ involvement or life-threatening) requiring treatment (BVAS score ≥ 3.0); The definition of severe illness is vasculitis with life-threatening or organ manifestations.
6. - for refractory LN

   * According to the 2019 American Society of Rheumatology (ACR) criteria, diagnosed with systemic lupus erythematosus, within 6 months prior to infusion, confirmed by renal tissue biopsy according to the 2003 International Society of Nephrology (ISN)/Society of Nephropathology (RPS) criteria as active, proliferative lupus nephritis (LN), type III or IV [excluding III (C), IV S (C), and IV G (C)], or type III/IV combined with type V, And have received standard treatment that is ineffective or relapses after disease remission. ②Positive anti-nuclear antibodies (ANA) and/or anti-dsDNA antibodies during the screening period. ③The SLE Disease Activity Index (SLEDAI-2000) score during the screening period is ≥ 8. SLEDAI-2000 clinical score ≥ 6 points, but low complement and/or anti ds-DNA positivity can be selected. ④The estimated survival period is at least 3 months.

Exclusion Criteria:

-Subjects who meet any of the following criteria should be excluded from this study:

1. Pregnant or lactating women;
2. If combined with alveolar hemorrhage, invasive pulmonary ventilation is required;
3. Refractory GPA and MPA: Combined with other autoimmune diseases involving multiple organ systems, such as EGPA, SLE, IgA vasculitis (Henoch Schönlein), rheumatoid arthritis, inflammatory myositis, anti-glomerular basement membrane disease, or cryoglobulinemia vasculitis;
4. Difficult to treat LN: severe extrarenal clinical manifestations such as lupus encephalopathy, pulmonary hemorrhage, lupus myocarditis, lupus enteritis, and lupus crisis; Other autoimmune diseases other than combined SLE, including dermatomyositis/polymyositis, mixed connective tissue disease, systemic sclerosis, rheumatoid arthritis, etc;
5. Individuals who are known to have allergic reactions, hypersensitivity reactions, intolerance, or contraindications to any component of PRG-1801 or drugs that may be used in the study (including fludarabine, cyclophosphamide, tocilizumab, albumin), or have experienced severe allergic reactions in the past;
6. A history of malignant tumors within 5 years (① subjects with cervical carcinoma in situ who have been completely removed and have not experienced recurrence or metastasis for at least 3 years may participate in this study. ② subjects with basal cell or squamous cell carcinoma who have been completely removed and have not experienced recurrence for at least 3 years may participate in this study);
7. Obvious evidence of cardiovascular disease as follows: a N-terminal B-type natriuretic peptide (NT proBNP)>8500ng/L; b. The New York Heart Association (NYHA) classifies heart failure as Grade IV; c. Patients who received hospitalization for unstable angina or myocardial infarction within 6 months prior to the first administration, or patients who received percutaneous cardiac intervention and received the most recent stent placement within 6 months or coronary artery bypass grafting within 6 months;
8. Received the following medication treatment within the prescribed time before single collection: ① Received B cell depletion therapy such as rituximab within 24 weeks; ② Received biological agents (such as TNF) within 4 weeks or 2 half-lives - Treatment with inhibitors, interleukin receptor inhibitors, belizumab, and tamoxifen; ③ Received treatment such as immunosuppressants within 2 weeks or 5 half-lives ; ④ If systemic glucocorticoids need to be used for a long time from 2 weeks before single collection to the study period, the dose of the hormone should not exceed 10mg/day; ⑤ Received plasma exchange or immunosorbent therapy within 24 weeks, and received intravenous immunoglobulin (IVIG) therapy within 4 weeks.
9. Vaccinate with live/attenuated vaccines within 4 weeks prior to single collection or during the study period;
10. Chronic and active hepatitis B ( the HBV DNA test is higher than 500IU/ml), hepatitis C (HCV), human immunodeficiency virus (HIV) infection, or syphilis infection;
11. There is an active infection that requires intravenous injection of antibiotics or hospitalization treatment;
12. Major surgery or surgical treatment caused by any reason within 4 weeks prior to enrollment;
13. Any serious and/or uncontrollable comorbidities that the researcher believes may interfere with the evaluation during the research process;
14. Participated in other intervention clinical trials within 3 months prior to enrollment or within 5 drug half-lives (whichever is longer);
15. Other conditions determined by the researcher as unsuitable for lymphocyte clearance or cell infusion, or other unsuitable patients for study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
AE Incidence of PRG-1801 Single Infusion | 24 months after PRG-1801 infusion
  AE Incidence of PRG-1801 Single Infusion
Types and incidence of dose-limiting toxicity(DLT) after PRG-1801 cells infusion in subjects with refractory ANCA-associated vasculitis and refractory LN. | 28 days and 3 months after PRG-1801 infusion
  To evaluate the DLT occurred within 28 days and 3 months after PRG-1801 infusion

SECONDARY OUTCOMES:
Therapeutic effects-For refractory ANCA-associated vasculitis(The proportion of subjects who maintained remission after cell infusion) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  The proportion of subjects who maintained remission after cell infusion
Therapeutic effects-For refractory ANCA-associated vasculitis(Changes in VDI (Vasculitis Damage Index) scores from baseline after cell infusion) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in VDI (Vasculitis Damage Index) scores from baseline after cell infusion
Therapeutic effects-For refractory ANCA-associated vasculitis (Changes in glomerular filtration rate compared to baseline after cell infusion in subjects with renal involvement.) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in glomerular filtration rate compared to baseline after cell infusion in subjects with renal involvement.
Therapeutic effects-For refractory LN (Changes in SLEDAI-2000 score from baseline after cell infusion) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in SLEDAI-2000 score from baseline after cell infusion
Therapeutic effects-For refractory LN (Changes in FACIT fatigue score from baseline after cell infusion ) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in FACIT fatigue score from baseline after cell infusion
Therapeutic effects-For refractory LN (Changes in PGA score (0-10) from baseline after cell infusion) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in PGA score (0-10) from baseline after cell infusion
Therapeutic effects-For refractory LN (Changes in eGFR(mL/min/1.73 m2) relative to baseline after cell infusion) | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in eGFR(mL/min/1.73 m2) relative to baseline after cell infusion
Therapeutic effects-For refractory LN (Changes in UPCR (g/24h）relative to baseline after cell infusion） | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  Changes in UPCR (g/24h）relative to baseline after cell infusion
Therapeutic effects-For refractory LN (The proportion of subjects who achieved overall response rate after cell infusion.） | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  The proportion of subjects who achieved overall response rate after cell infusion.
Therapeutic effects-For refractory LN（The proportion of subjects who achieved complete renal response after cell infusion.） | Month1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  The proportion of subjects who achieved complete renal response after cell infusion.
PK feature evaluation (PK parameters related to CAR copy number） | baseline, Day2, Day6, Day10, Day21, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 after cell infusion
  PK parameters related to CAR copy number
Serum sBCMA level | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum sBCMA level (count/uL)
Serum ANCA titer level (AAV) | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum ANCA titer level (AAV)
Serum dsDNA level (LN) | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum dsDNA level (IU/mL)
Serum ANA titer level (LN) | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum ANA titer level (IU/mL)
Serum complement C3 levels | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum complement C3 levels (g/L)
Serum complement C4 levels | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum complement C4 levels (g/L)
Serum immunoglobulin quantification | baseline, Day14, Day28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24 month after cell infusion
  Serum immunoglobulin quantification (g/L)
Levels of CRP levels | baseline, Day2, Day6, Day10, Day14, Day21, Day28 after cell infusion
  Levels of CRP levels (mg/L)
Levels of ferritin levels | baseline, Day2, Day6, Day10, Day14, Day21, Day28 after cell infusion
  Levels of ferritin levels (ug/L)
Levels of cytokine levels | baseline, Day2, Day6, Day10, Day14, Day21, Day28 after cell infusion
  Levels of cytokine levels (pg/mL)
Changes of peripheral blood lymphocyte subsets | baseline, Day2, Day6, Day10, Day14, Day21, Day28, Month 2, Month 3, Month 6 after cell infusion
  Changes of peripheral blood lymphocyte subsets (count/uL)
Expression levels of BCMA on peripheral blood B cell subsets surface | baseline, through study completion, an average of 2 years
  Expression levels of BCMA on peripheral blood B cell subsets surface (%), using flow cytometer method.
The level of anti drug antibody (ADA) | baseline, through study completion, an average of 2 years
  The level of anti drug antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Lingli Dong, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No